CLINICAL TRIAL: NCT03418259
Title: Study of Patients With Dry Eyes, Keratoconjunctivitis Sicca, During Treatment With Intra-Nasal Mechanical Stimulation (INMEST)
Brief Title: Intra-Nasal Mechanical Stimulation (INMEST) as a Treatment of Keratoconjunctivitis Sicca (Dry Eye Syndrome)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Källmark Clinic (Other)
Responsible Party: Principal Investigator, Jan-Erik Juto, Principal Investigator, M.D., Ph.D., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INMESTfordryeyes2018
Record Dates: First submitted 2018-01-19; First posted 2018-02-01 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Keratoconjunctivitis Sicca (KCS)
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Intervention Model Description: Double blinded randomised clinical trial
Who Masked: Participant, Investigator
Masking Description: Placebo device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active KCS Medical Device (Experimental)
  Interventions: Device: KCS Medical Device
- Inactive KCS Medical Device (Placebo Comparator)
  Interventions: Device: KCS Medical Device

INTERVENTIONS:
Device: KCS Medical Device — Patient treated 6 times with the Active KCS Medical Device during 2 weeks.
  Arms: Active KCS Medical Device
Device: KCS Medical Device — Patient treated 6 times with the Inactive KCS Medical Device during 2 weeks.
  Arms: Inactive KCS Medical Device

SUMMARY:
The purpose of the study is to evaluate how treatment with Intra-Nasal Mechanical Stimulation (INMEST) in the nasal cavity in patients with Keratoconjunctivitis sicca can relieve these symtoms.

ELIGIBILITY:
Inclusion Criteria:

* Ocular surface disease index, OSDI > 12 points.
* Non-invasive breakup time, NIBUT < 11 seconds.

Exclusion Criteria:

* Ocular surface disease index, OSDI < 12 points.
* Non-invasive breakup time, NIBUT > 11 seconds.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Ocular surface disease index, OSDI | Change from Baseline Ocular surface disease index at two weeks.
  12-item scale for the assessment of symptoms related to dry eye disease and their effect on vision. Scale 0-100, normal value range 0-12.

SECONDARY OUTCOMES:
Noninvasive breakup time, NIBUT | Change from Baseline Noninvasive breakup time at two weeks.
  Assessment of tear film stability. Normal value at least 11 seconds.
Meibography | Change from Baseline Meibo scale value at two weeks.
  Imaging study method for directly visualizing the morphology of Meibomian glands in vivo. Fat amount in the Meibomian glands is quantified and stated in percent. A Meibo scale value over 25 % is considered abnormal.
Phenol Red Thread Test, PRT | Change from Baseline lacrimation assessed with Phenol Red Thread Test value at two weeks.
  Measurement of lacrimation, stated in millimetres. Normal value is 12-20 millimetres.
Tear (lacrimal) meniscus height | Change from Baseline Tear (lacrimal) meniscus height at two weeks.
  Tear meniscus height measured medially on the lower eyelid. Stated in millimetres. Normal value is over 0,2 mm.
Lissamin green test | Change from Baseline spread of dry cell patches quantified with Lissamin green test at two weeks.
  A strip of paper containing lissamine green is diluted with saline, and then dropped into the eye. The colour of the paper will disclose any dry cell patches in the eye.
Corneal staining with fluorescein | Change from Baseline Efron Grading Scale value at two weeks.
  Fluorescein is used to describe the severity of damaged epithelial cells on cornea. Efron Grading Scale, 1-5. 0 is normal value.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Erik Juto, M.D., Ph.D., Principal Investigator — Department of Clinical Science, Intervention and Technology (CLINTEC), H9, Karolinska Institutet
Locations (1):
- Källmarkskliniken, Stockholm, Sweden